CLINICAL TRIAL: NCT06960980
Title: Improving ADHD Teen Driving - Virtual Reality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0273; R01HD084430-06A1 (NIH)
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Visual attention; Automobile Driving
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FOCAL+ Training (Experimental): Enhanced FOcused Concentration and Attention Learning driver training using desktop computer and fixed base driving simulator
  Interventions: Behavioral: FOCAL+
- Virtual Reality - FOCAL+ (Experimental): Enhanced FOcused Concentration and Attention Learning driver training using virtual reality
  Interventions: Behavioral: VR-FOCAL+
- Wait-list Control (No Intervention): Teens will wait approximately 1 year to receive FOCAL+ training. In order to control for experience with the driving simulator across groups, teens in this group will attend 5 weekly sessions where they will experience five 5-minute drives in the driving simulator. During the drives, teens will be cued to a complete a visual search task which will require them to divert their gaze from the road. Teens in this group will not receive feedback regarding eye glances during these drives.

INTERVENTIONS:
Behavioral: FOCAL+ — Weekly for 5 weeks, teens complete a computer training program designed to train teens to limit the length of glances away from the roadway. During phase 1 of each training session, on a computer, the top portion of the screen plays a simulated video drive while the bottom half of the screen contains a map. Teens complete tasks that require switching between the 2 halves of the screen. While doing so, they receive feedback regarding how long they are looking away from the driving portion of the screen. During phase 2 of each training session, teens will complete five 5-minute simulated drives using a fixed-base driving simulator. During the drives, teens will be cued to a complete a visual search task which will require them to divert their gaze from the road. Eye tracking goggles will monitor eye glances and provide real time auditory feedback when a visual glance away from the roadway exceeds 2 secs.
  Arms: FOCAL+ Training
Behavioral: VR-FOCAL+ — Weekly for 5 weeks, teens complete a training program designed to train teens to limit the length of glances away from the roadway. The training has two phases, each of which will be administered using immersive virtual reality. The first phase will have teens switch between the upper half of a virtual reality screen which will play a simulated video drive while the bottom half contains a map. Teens complete tasks that require switching between the 2 halves of the screen. While doing so, they receive feedback regarding how long they are looking away from the driving portion of the screen. During the second phase of each session, teens will complete five 5-minute simulated drives in a virtual reality environment where teens will be cued to a complete a visual search task which will require them to divert their gaze from the road. Eye tracking will monitor eye glances and provide real time auditory feedback when a visual glance away from the roadway exceeds 2 secs.
  Arms: Virtual Reality - FOCAL+

SUMMARY:
Teens with Attention-Deficit/Hyperactivity Disorder (ADHD) have high rates of negative driving outcomes, including motor vehicle crashes, which may be caused by visual inattention (i.e., looking away from the roadway to perform secondary tasks). Two versions of a driving intervention that trains teens to reduce instances of looking away from the roadway will be tested in teens with ADHD.

DETAILED DESCRIPTION:
Motor vehicle crashes (MVC) are the leading causes of death among teens with eight teens dying per day in an MVC. Teens with Attention-Deficit Hyperactivity Disorder (ADHD) are at twice the risk of MVC compared to teen drivers without ADHD. A programmatic line of research by this investigative team has identified long (>2 secs) glances away from the roadway, particularly during engagement with secondary tasks, as being a key mechanism in ADHD teen driving risk. In the original research grant, the investigative team developed and tested a driver training program, enhanced FOcused Concentration and Attention Learning (FOCAL+), to specifically target reducing rates of extended glances away from the roadway in teens with ADHD. In a randomized controlled trial (RCT), teens with ADHD randomly assigned to FOCAL+ demonstrated 41% fewer long-glances and less variability in lane position during simulated driving assessments conducted immediately after the final training session, and 1- and 6-months post-training compared to teens assigned to modified driver's training. Moreover, during naturalistic driving over the course of a year of driving, FOCAL+ teens had 40% less risk of a crash/near-crash event than control teens. However, there are considerable barriers to disseminating FOCAL+ in its current format. FOCAL+, as implemented in the RCT, requires costly (~$90K) hardware and software that are quite complex to use. Though there has been much interest in offering this training since publication of our RCT results, key stakeholders have reported that the expense and complexity of the hardware and software requirements are barriers to adoption. In the proposed study, with input from relevant stakeholders, FOCAL+ training will be converted to an immersive virtual reality (iVR) platform. iVR-FOCAL+ will provide an affordable ($5K), single hardware, single software, easily-executable solution that implementation sites (i.e., driving schools, outpatient occupational therapy) will be able to afford, adopt, and offer to teens with ADHD. Using a hybrid effectiveness-implementation design, teens with ADHD will be randomly assigned to receive either iVR-FOCAL+, the original FOCAL+ or a wait-list control group. The iVR-FOCAL+ training will be implemented in real-world, non-research settings (i.e., driving schools, outpatient occupational therapy). At baseline and 1- and 6-months post-training, teens' driving skills will be assessed during driving simulation. Naturalistic driving will be assessed during the year after training using video event recorders installed in the teen's car. Training costs and implementation outcomes (e.g., barriers to implementation) for each training will be collected. Using these data, the investigators will examine the relative effectiveness and cost-effectiveness of iVR-FOCAL+ intervention compared to FOCAL+ training. Finally, implementation of iVR-FOCAL+ will be described. The proposed research has the potential to facilitate adoption and eventual dissemination of a training program that can prevent injuries and fatalities among a high-risk population of teens as well as among those who share their roadways.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16-19.
2. Teens will meet DSM ADHD criteria for ADHD-Predominantly Inattentive Presentation or ADHD-Combined Presentation based on the K-SADS interview.
3. Possess a valid driver's license and regularly spend at least 3 hours per week engaged in unsupervised driving.
4. IQ ≥80 as measured by the Kauffman Brief Intelligence Scale - Second Edition (KBIT-2).
5. Parent willing to participate.

Exclusion Criteria:

1. On ADHD medication that cannot be washed out on assessment days.
2. Drug or alcohol dependence based on self-report on the Simple Screening Instrument for Alcohol and Other Drugs survey.
3. On psychotropic or neuroleptic medications.
4. At-risk for motion sickness in the driving simulator or in virtual reality.
5. History of moderate to severe head trauma, neurological disorder, or any other organic disorder that could possibly affect brain function.
6. Cannot see the secondary task stimuli without the use of glasses (contacts acceptable).

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of extended glances away from the roadway during simulated driving | 1-month post-training
  Participants will complete a simulated drive in a driving simulator with an integrated eye-tracking system. Participants will complete two 15-minute drives. During each drive, participants will engage in 14 secondary tasks. The secondary task consist of searching for streets on a GPS map for 20 seconds. Eye gaze will be sampled continuously. Eye gaze data will be summarized by calculating the number of extended (≥2 secs) glances away from the roadway during the 14 secondary task periods per drive. Descriptive estimates will reflect averages across the 2 drives. However, for analyses, estimates for each drive will be statistically modeled with a two-level drive variable.
Number of extended glances away from the roadway during simulated driving | 6-months post-training
  Participants will complete a simulated drive in a driving simulator with an integrated eye-tracking system. Participants will complete two 15-minute drives. During each drive, participants will engage in 14 secondary tasks. The secondary task consist of searching for streets on a GPS map for 20 seconds. Eye gaze will be sampled continuously. Eye gaze data will be summarized by calculating the number of extended (≥2 secs) glances away from the roadway during the 14 secondary task periods per drive. Descriptive estimates will reflect averages across the 2 drives. However, for analyses, estimates for each drive will be statistically modeled with a two-level drive variable.

SECONDARY OUTCOMES:
Standard Deviation of Lateral Position during simulated driving | 1-month post-training
  Participants will complete a simulated drive in a driving simulator with an integrated eye-tracking system. Participants will complete two 15-minute drives. During each drive, participants will engage in 14 secondary tasks. The secondary task consist of searching for streets on a GPS map for 20 seconds. Lateral position will be sampled continuously. Standard deviation of lane position will be calculated for the 14 secondary task periods per drive. Estimates will reflect averages across the 2 drives. However, for analyses, estimates for each drive will be statistically modeled with a two-level drive variable.
Standard Deviation of Lateral Position during simulated driving | 6-months post-training
  Participants will complete a simulated drive in a driving simulator with an integrated eye-tracking system. Participants will complete two 15-minute drives. During each drive, participants will engage in 14 secondary tasks. The secondary task consist of searching for streets on a GPS map for 20 seconds. Lateral position will be sampled continuously. Standard deviation of lane position will be calculated for the 14 secondary task periods per drive. Estimates will reflect averages across the 2 drives. However, for analyses, estimates for each drive will be statistically modeled with a two-level drive variable.

OTHER OUTCOMES:
Rate of crashes and near-crashes recorded with DriveCam | 12-months post-training
  DriveCam is an event-triggered device with a pair of cameras that are mounted to the rear view mirror of the participant's car. The device has a forward-road facing camera and another camera that faces the driver. Both cameras continuously record but only save to memory when a built-in accelerometer exceeds a set g force threshold. Any g-force event that exceeds .6 g-force will be coded using codings of crashes (i.e., collision with another vehicle or object) or near-crashes (i.e., an evasive maneuver performed to avoid a MVC). This outcome will include the rate of crashes or near-crashes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff N Epstein, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical data that will be preserved and shared are demographic data, diagnostic data and intelligence testing results, among other data pertinent to the study. Research data that will be shared include the driving history, driving simulation, eyetracking data, and driving event codings.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study team will submit an initial batch of processed and cleaned data to the NICHD Data and Specimen Hub (DASH) after the first 50 participants have been enrolled in order to develop a pipeline for submitting study data to DASH. Along with these data, the investigators will develop and submit any data dictionaries and codebooks for these data. All remaining data will be submitted within 1 year of the last patient's last study visit, 4 months prior to any publication date, or 6 months before the end of the performance period, whichever is sooner.
Access Criteria: Clinical data will be shared with controlled access in NICHD Data and Specimen Hub (DASH) for general research use, as allowed by the participant's informed consents and the institutional certification. To access study data within DASH, users must submit a Data Request Checklist to DASH, sign the NICHD DASH Data Use Agreement, and submit proof of IRB approval.

REFERENCES:
- [Background] Epstein JN, Garner AA, Kiefer AW, Peugh J, Tamm L, MacPherson RP, Simon JO, Fisher DL. Trial of Training to Reduce Driver Inattention in Teens with ADHD. N Engl J Med. 2022 Dec 1;387(22):2056-2066. doi: 10.1056/NEJMoa2204783. PMID 36449421